CLINICAL TRIAL: NCT05320120
Title: Investigation of Intranasal Ketamine Related Changes in Attentional Brain Networks With Functional and Structural MRI: a Placebo Controlled, Randomized, Cross-over Trial
Brief Title: Investigation of Intranasal Ketamine Related Changes in Attentional Brain Networks With Functional and Structural MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rupert Lanzenberger (Other)
Responsible Party: Sponsor-Investigator, Rupert Lanzenberger, Prof. Dr. Rupert Lanzenberger, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PSY-NIL-0011
Record Dates: First submitted 2022-02-28; First posted 2022-04-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Ketamine Treatment
MeSH Terms: interventions — Esketamine; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first 56mg esketamine (2x Spravato® 28 mg nasal spray), then placebo (Experimental)
  Interventions: Drug: 56mg esketamine (2x Spravato® 28 mg nasal spray); Drug: 0.9% saline solution nasal spray
- first placebo (0.9% saline solution nasal spray), then ketamine (Experimental)
  Interventions: Drug: 56mg esketamine (2x Spravato® 28 mg nasal spray); Drug: 0.9% saline solution nasal spray

INTERVENTIONS:
Drug: 56mg esketamine (2x Spravato® 28 mg nasal spray) — 56mg esketamine (2x Spravato® 28 mg nasal spray)
Drug: 0.9% saline solution nasal spray — 0.9% saline solution nasal spray

SUMMARY:
Subanesthetic ketamine is currently used as a rapid-acting antidepressant. It is an antagonist of the N-methyl-d-aspartate (NMDA) receptor, but former results indicate that its action also depends on the noradrenaline system and the locus coeruleus (LC).

Based on this known impact of ketamine on the sympathetic nervous system the aim of this study is to investigate the effects of intranasal esketamine on LC related attentional brain networks in task based functional MRI, to relate those attention network changes to behavioural measures and to predict ketamine related attention network changes by brain structure.

ELIGIBILITY:
Inclusion Criteria:

* General health (no serious internal or neurologic pre-existing conditions) based on medical history, physical examination and structured clinical interview for DSM-IV (SCID)
* Age 18 to 55 years
* Right-handedness (due to potential lateralization effects of left-handed subjects)
* Willingness and competence to sign the informed consent form

Exclusion Criteria:

* Current or history of psychiatric or neurological disease
* Current medical illness requiring treatment
* Current or former substance abuse
* Pregnancy or current breastfeeding
* Diagnosis of an Axis-1 psychotic disorder in a first-degree relative
* Known aneurysmal vascular disease based on medical history (including intracranial, thoracic, or abdominal aorta, or peripheral arterial vessels), history of intracerebral haemorrhage, recent (within 6weeks) cardiovascular event, including myocardial infarction (MI)
* Significant pulmonary insufficiency, including COPD; sleep apnoea with morbid obesity (BMI ≥35), uncontrolled brady- or tachyarrhythmias that lead to haemodynamic instability; history of an MI, haemodynamically significant valvular heart disease or heart failure (NYHA Class III-IV)
* Hyperthyroidism that has not been sufficiently treated
* History of brain injury, hypertensive encephalopathy, intrathecal therapy with ventricular shunts, or any other condition associated with increased intracranial pressure
* Child-Pugh class C (severe) hepatic impairment
* Any contraindication for MRI (e.g., MR incompatible implants, etc.) including dental implants causing signal artifacts
* Failure to comply with the study protocol or to follow the instruction of the investigating team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
BOLD response assessed with fMRI to arousal task | up to two weeks
  Blood oxygen level (BOLD) response assessed with functional magnetic resonance imaging (fMRI) during an arousal task

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Vienna, Austria